CLINICAL TRIAL: NCT04138615
Title: Analgesics in the Pre-hospital Setting: Implications on Hemorrhage Tolerance - Morphine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU 092017-070
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine (Experimental): Morphine will be administered intravenously
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Saline will be administered intravenously
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Morphine — Subjects will receive Morphine while the effects of this drug on tolerance to a hemorrhagic insult will be assessed.
  Arms: Morphine
Other: Placebo — Subjects will receive saline while the effects of this drug on tolerance to a hemorrhagic insult will be assessed.
  Arms: Placebo

SUMMARY:
We are examining how morphine (a commonly used pain medication) will alter responses to simulated blood loss in humans. To simulate blood loss in our research laboratory, participants will complete a test with their lower body in a custom-designed vacuum chamber for a brief period of time.

DETAILED DESCRIPTION:
Pain management on the battlefield is critical for the wellbeing of the soldier. Given that a hemorrhagic injury on the battlefield is virtually always associated with pain, it is paramount that the selected pain medication does not disrupt appropriate physiological mechanisms that are beneficial towards the maintenance of blood pressure and vital organ blood flow during that hemorrhagic insult. Current guidelines for the selection of pain medications of a hemorrhaging soldier are based upon limited scientific evidence, with the vast majority of supporting studies being conducted on anesthetized animals. Thus, the interaction between hemorrhagic shock and pain medications commonly employed on the battlefield is yet to be determined in the conscious humans.

With this background, we will test the hypothesis that morphine will impair the capacity for a conscious human to tolerate a hemorrhagic insult.

The obtained data will provide the necessary scientific evidence in humans to support the Committee on Tactical Combat Casualty Care (CoTCCC) guidelines on the analgesic of choice for moderate to severe injuries where the casualty is in hemorrhagic shock. Notably, such data will identify the analgesic that least compromises a human's ability to tolerate a hemorrhagic insult, ultimately providing critical information to the combat medic on which analgesic should be employed for such an injury.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-obese (body mass index less than 30 kg/m2)
* Body mass greater than or equal to 65 kg

Exclusion Criteria:

* Subjects who have cardiac, respiratory, neurological and/or metabolic illnesses
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy or breast feeding
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Positive urine drug screen
* Currently taking pain modifying medication(s)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine First, Then Placebo: Morphine will be administered first, followed by the Placebo (saline) visit.
- Placebo First, Then Morphine: Placebo visit (saline) first, then Morphine visit
Period: Overall Study
Arm/Group | Morphine First, Then Placebo | Placebo First, Then Morphine
Started | 19 | 25
Completed | 14 | 16
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- All Participants: These numbers are for all participants
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Tolerance to Simulated Hemorrhage
Description: Tolerance to a simulated hemorrhagic challenge will be assessed, for both the placebo and morphine limbs, by causing progressive central hypovolemia via lower-body negative pressure (LBNP). This progressive LBNP challenge will be performed until the onset of syncopal symptoms (defined as: profound bradycardia, a precipitous drop in arterial blood pressure and accompanying narrowing of pulse pressure, a sustained systolic blood pressure less than 80 mmHg, and/or subjective symptoms such as light-headedness, sweating, nausea, or dizziness). The primary variable will be the quantification of LBNP that is required to cause these symptoms. This quantification will be objectively measured via a cumulative stress index which is calculated as the sum of the product of the LBNP level and the duration of each level, until test termination (i.e., 40 mmHg x 3 min + 50 mmHg x 3 min, etc). A larger cumulative stress index represents a greater tolerance
Time Frame: 30 minutes from the onset of applying lower-body negative pressure
Measure: Median (Inter-Quartile Range); unit: CSI: Cumulative Stress Index
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 30 | 30
CSI: Cumulative Stress Index | 385 [251 to 728] | 692 [473 to 997]

2. Secondary Outcome: Pain Assessment - Algometer
Description: Pain assessments will be conducted using a digital algometer to obtain maximum pain thresholds caused by pressure. This pain assessment technique is conducted by applying the tip of a hand-held digital algometer on the subject's digit. Force is gradually increased and the peak force is recorded when the subject first reports a painful sensation. Removal of the pressure from the algometer immediately relieves the painful sensation and the subject can voluntarily stop the test at any time. This assessment will be performed when the subject has received placebo and morphine.
Time Frame: 30 minutes from the onset of the protocol
Measure: Median (Inter-Quartile Range); unit: Kilogram force/0.13 cm^2
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 30 | 30
Kilogram force/0.13 cm^2 | 1.1 [0.9 to 1.5] | 0.9 [0.7 to 1.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from until discharge from the final data collection visit, which typically occurred 6 to 12 months after consent/screening.
Description: Each participant completed both drug and placebo conditions, therefore, groups are combined for adverse event reporting.
Groups:
- Placebo Trial; Morphine Trial: These numbers are for all participants
Arm/Group | Placebo Trial | Morphine Trial
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04138615/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT04138615/ICF_003.pdf